CLINICAL TRIAL: NCT00313261
Title: An Open-Label, Phase II Study to Evaluate Safety, Tolerability, Antiviral Activity and Biochemical and Immunological Responses of L-FMAU (Clevudine) in Chronic Hepatitis B Patients of L-FMAU-201 Placebo Group
Brief Title: Safety and Efficacy Study of L-FMAU in Chronic HBV Patients of L-FMAU-201 Placebo Group
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bukwang Pharmaceutical (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-FMAU-203
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — clevudine

INTERVENTIONS:
Drug: Clevudine

SUMMARY:
The purpose of this study is to evaluate the safety and antiviral activity of clevudine 30 mg QD for treatment of longer period (24 weeks) in patients chronically infected with HBV.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received placebo in L-FMAU-201 study
2. Female of childbearing potential with a negative serum (beta-HCG) pregnancy test within 14 days of starting therapy.
3. Patients who were able to give written informed consent prior to study start and to comply with the study requirements.
4. Patients who met the following criteria after completion of the Week 48 visit were to have additional follow-up visits at Weeks 54 and 60:

1)had received no additional therapy since completion of 24-week treatment of clevudine and 2)experienced a >= 1 log10 decrease from baseline in HBV DNA at Week 48

Exclusion Criteria:

1. Patient with HBeAg seroconverted to anti-HBe at the last 2 consecutive visits (one month apart) in L-FMAU-201 study.
2. Patient who was currently receiving antiviral, immunomodulatory or corticosteroid therapy.
3. Patient who was treated with lamivudine, lobucavir, famciclovir, adefovir or any other investigational nucleoside for HBV infection after cessation of treatment in L-FMAU-201 study.
4. Patient who had a history of ascites, variceal hemorrhage or hepatic encephalopathy.
5. Patient who was co-infected with HCV, HDV or HIV.
6. Patient with clinical evidence of cirrhosis or hepatocellular carcinoma (®-Fetoprotein)Evaluation was based on alpha-fetoprotein primarily. If alpha-fetoprotein level was suggestive of cirrhosis or hepatocellular carcinoma, confirmation was made with ultrasonography etc.
7. Patient who was pregnant or breast-feeding.
8. Patient who was unwilling to use an "effective" method of contraception during treatment period and for up to 3 months after cessation of therapy. For males, condoms should be used. Females must be surgically sterile (via hysterectomy or bilateral tubal ligation), post-menopausal or using at least a medically acceptable barrier method of contraception (i.e., IUD, barrier methods with supermicide or abstinence)
9. Patient who had a clinically relevant history of abuse of alcohol or drugs.
10. Patient who had a significant gastrointestinal, renal, hepatic (decompensated), bronchopulmonary, neurological, cardiovascular, oncologic or allergic disease.
11. Patient who had creatinine clearance less than 60mL/min as estimated by the following formula:

(140-age in years) (body weight [kg])/(72) (serum creatinine [mg/dL]) [Note: multiply estimates by 0.85 for women]

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-06; Study Completion 2005-02

PRIMARY OUTCOMES:
Efficacy: Change from baseline in HBV DNA (log10)
Safety: Laboratory tests, Adverse Events, Vital Signs, ECG

SECONDARY OUTCOMES:
Efficacy
Proportion of patients with HBV DNA below the assay Limit of Detection (4,700 copies/mL by Digene Hybrid Capture II)
Biochemical improvement (ALT normalization)
Serology Proportion of patients with HBeAg loss Seroconversion rate (HBeAg loss and anti-HBe gain)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Suk Lee, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (7):
- South Korea (7):
  - Korea University Guro Hospital, Guro-dong, Guro-ku, Seoul
  - Seoul National University, Yeongeon-dong, Jongno-Gu, Seoul
  - Samsung Medical Center, Ilwon-dong, Kangnam-Gu, Seoul
  - Yongdong Severance Hospital, Togok-tong, Kangnam-Gu, Seoul
  - Asan Medical Center, P’ungnabi-dong, Songpa-Gu, Seoul
  - Ewha Womans University Hospital, Mokdong, Yangchon-Gu, Seoul
  - St. Mary's Hospital, Youido, Yougdungpo-Gu, Seoul